CLINICAL TRIAL: NCT04591548
Title: Biomarkers in Endometriosis
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Vid Jansa, Principal Investigator, University Medical Centre Ljubljana
Other Study IDs: BEND
Record Dates: First submitted 2020-08-01; First posted 2020-10-19 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Endometriosis
Keywords: Endometriosis; Biomarkers
MeSH Terms: conditions — Endometriosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — peritoneal fluid precipitate, serum precipitate, uterine fluid precipitate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis: All patients had laparoscopy due to infertility (and endometriosis). All women had BMI in normal range and regular menstrual cycle (21-35 days). Partner's semen analysis was normal in all cases. The investigators excluded patients with hormonal therapy in the last year, irregular menstrual cycle, smokers and patients with autoimmune diseases, malignant or suspected malignant diseases, previous pelvic inflammatory disease, leiomyoma uteri or polycystic ovaries. None of the patients had previous pelvic surgery.
  Interventions: Diagnostic Test: proteomic analyses, ELISA validation of peritoneal fluid, blood and uterine fluid sample
- Primary infertility: All patients had laparoscopy due to infertility (and endometriosis). All women had BMI in normal range and regular menstrual cycle (21-35 days). Partner's semen analysis was normal in all cases. The investigators excluded patients with hormonal therapy in the last year, irregular menstrual cycle, smokers and patients with autoimmune diseases, malignant or suspected malignant diseases, previous pelvic inflammatory disease, leiomyoma uteri or polycystic ovaries. None of the patients had previous pelvic surgery.
  Interventions: Diagnostic Test: proteomic analyses, ELISA validation of peritoneal fluid, blood and uterine fluid sample

INTERVENTIONS:
Diagnostic Test: proteomic analyses, ELISA validation of peritoneal fluid, blood and uterine fluid sample — All samples were collected during laparoscopy, before any intraabdominal procedure was done. Indication for surgery was clinical (not for research purpose). All sample collection procedures was mimic regular clinical procedures.

SUMMARY:
Endometriosis is a common gynecological benign disease which significantly compromise quality of life in patients and is a major cofactor of infertility. With the proteomic approach the investigators will search for proteins with significantly different levels in peritoneal fluid, serum and uterine fluid samples of women with endometriosis versus control group. Results will be validate using ELISA aproach.

DETAILED DESCRIPTION:
Informed consent will be obtained from all individual participants included in the study. Blood sample will be obtained the day before laparoscopic surgery during regular clinical preoperative procedures. Peritoneal fluid and uterine fluid will be obtained during regular laparoscopic procedure indicated for infertility, the exact protocol of sample obtaining will be revealed after publication of results. The aim of the study was to identify potential diagnostic and predictive biomarkers or drug targets.

ELIGIBILITY:
Inclusion Criteria:

* primary infertility
* normal semen analysis of the partner
* normal BMI.

Exclusion Criteria:

* hormonal therapy in the last year,
* irregular menstrual cycle,
* previous pelvic surgery,
* history of previous pelvic inflammatory disease,
* smokers and patients with autoimmune diseases,
* malignant or suspected malignant diseases,
* previous pelvic inflammatory disease, leiomyoma uteri or polycystic ovaries

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gynecological condition
Study Population: Patients with primary infertility or endometriosis with clinical indication for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Derivation of the panel of proteins indicative of endometriosis using comparative proteomics | 3 years to collect all speciments
  The aim of the study is to identify proteins with different levels in cases versus controls these proteins could be new candidates for biomarkers of endometriosis. Differentially expressed proteins are candidates for diagnostic and predictive biomarkers. To identify differentially expresed proteins in discovery phase of the study proteomic aproach will be used.

SECONDARY OUTCOMES:
Concentrations of proteins in body fluids to validate the identified panel of proteins indicative of endometriosis | 3 years to collect all speciments
  Using pairs of subjects with and without endometriosis, the derivation of the panel of proteins in body fluids (peritoneal fluid, peripheral blood, uterine fluid samples) gathered through proteomic aproach will be validated using ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Vid Jansa, MD, Principal Investigator — UKCLjubljana

IPD SHARING:
Plan to Share IPD: No